CLINICAL TRIAL: NCT03381274
Title: A Multiarm, Open-label, Multicenter, Phase 1b/2 Study to Evaluate Novel Combination Therapies in Subjects With Previously Treated Advanced EGFRm NSCLC
Brief Title: Oleclumab (MEDI9447) Epidermal Growth Factor Receptor Mutant (EGFRm) Non-small Cell Lung Cancer (NSCLC) Novel Combination Study
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6070C00004
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: EGFR mutated; CD73; A2AR; Oleclumab; MEDI9447; AZD4635; Osimertinib; NSCLC; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Oleclumab Dose 1 + Osimertinib Dose 1 (Experimental): In Part 1 (dose-escalation), participants will receive intravenous oleclumab (MEDI9447) Dose 1 every 2 weeks (Q2W) and oral osimertinib Dose 1 once daily (QD).
  Interventions: Biological: Oleclumab; Drug: Osimertinib
- Oleclumab Dose 2 + Osimertinib Dose 1 (Experimental): In Part 1 (dose-escalation), participants will receive intravenous oleclumab Dose 2 Q2W and oral osimertinib Dose 1 QD. In Part 2 (dose-expansion), participants (including participants dosed at the RP2D in Part 1) will receive IV oleclumab Dose 2 Q2W and oral osimertinib Dose 1 QD until documentation of disease progression, intolerable toxicity, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Biological: Oleclumab; Drug: Osimertinib
- Oleclumab Dose 1 + AZD4635 Dose 1 (Experimental): In Part 1 (dose-escalation), participants will receive intravenous oleclumab Dose 1 Q2W and oral AZD4635 Dose 1 QD.
  Interventions: Biological: Oleclumab; Drug: AZD4635
- Oleclumab Dose 1 + AZD4635 Dose 2 (Experimental): In Part 1 (dose-escalation), participants will receive intravenous oleclumab Dose 1 Q2W and oral AZD4635 Dose 2 QD.
  Interventions: Biological: Oleclumab; Drug: AZD4635
- Oleclumab Dose 2 + AZD4635 Dose 2 (Experimental): In Part 1 (dose-escalation), participants will receive intravenous oleclumab Dose 2 Q2W and oral AZD4635 Dose 2 QD.
  Interventions: Biological: Oleclumab; Drug: AZD4635

INTERVENTIONS:
Biological: Oleclumab — Participants will receive oleclumab in combination with osimertinib or AZD4635 as stated in the arms' description.
  Other Names: MEDI9447
Drug: Osimertinib — Participants will receive osimertinib in combination with oleclumab as stated in the arms' description.
  Other Names: Tagrisso®
  Arms: Oleclumab Dose 1 + Osimertinib Dose 1; Oleclumab Dose 2 + Osimertinib Dose 1
Drug: AZD4635 — Participants will receive AZD4635 in combination with oleclumab as stated in the arms' description.
  Arms: Oleclumab Dose 1 + AZD4635 Dose 1; Oleclumab Dose 1 + AZD4635 Dose 2; Oleclumab Dose 2 + AZD4635 Dose 2

SUMMARY:
The objective of this study is to investigate the safety, tolerability, and antitumor activity of novel combination therapies administered in participants with advanced EGFRm NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
3. Weight ≥ 35 kg
4. Diagnosed with histologically or cytologically confirmed locally advanced/metastatic NSCLC with EGFRm

   * For Arm A (Oleclumab + Osimertinib arms): must have received 1 prior line of therapy with an EGFR tyrosine kinase inhibitor (TKI) and confirmed T790M negative
   * For Arm B (Oleclumab + AZD4635 arms): must have received at least 2 but not more than 4 prior lines of therapy.

Exclusion Criteria:

1. Receipt of an EGFR TKI within 14 days of the first dose of study treatment
2. Receipt of any conventional or investigational anticancer therapy not otherwise specified within 21 days of the planned first dose
3. Prior receipt of any investigational immunotherapy. Participants may have received agents that have local health authority approval for the disease indication
4. Concurrent enrollment in another therapeutic clinical study. Enrollment in observational studies will be allowed.
5. Participants with a history of venous thrombosis within the past 3 months
6. Participants with prior history of myocardial infarction, transient ischemic attack, or stroke in the last 6 months
7. Active or prior documented autoimmune or inflammatory disorders within the past 3 years prior to the start of treatment
8. Other invasive malignancy within 2 years
9. Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression
10. Current or prior use of immunosuppressive medication within 14 days prior to the first dose

Additional Exclusion Criteria for Arm A

1. Concurrent treatment (or inability to stop therapy) with medications or herbal supplements known to be potent inducers of cytochrome P (CYP) 3A4
2. Participants has a history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD
3. Participants requires continuous supplemental oxygen for any reason

Additional Exclusion Criteria for Arm B

1. Herbal preparations/medications are not allowed throughout the study
2. History of seizures excluding those that occurred due to previously untreated CNS metastasis

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2026-04-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (11):
- United States (9):
  - Research Site, La Jolla, California
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- Research Site, Seoul, South Korea
- Research Site, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Kim DW, Kim SW, Camidge DR, Shu CA, Marrone KA, Le X, Blakely CM, Park K, Chang GC, Patel SP, Kar G, Cooper ZA, Samadani R, Pluta M, Kumar R, Ramalingam S. CD73 Inhibitor Oleclumab Plus Osimertinib in Previously Treated Patients With Advanced T790M-Negative EGFR-Mutated NSCLC: A Brief Report. J Thorac Oncol. 2023 May;18(5):650-656. doi: 10.1016/j.jtho.2022.12.021. Epub 2023 Jan 11. PMID 36641093
- See also: D6070C00004 redacted protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6070C00004&attachmentIdentifier=f05a0e14-fcde-4156-bdf4-8f6c64c7e249&fileName=protocol-d6070c00004-amendment-4-Redacted_18May2022.pdf&versionIdentifier=
- See also: D6070C00004 SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6070C00004&attachmentIdentifier=3142be22-09f6-4179-9790-abf963256362&fileName=d6070c00004-sap-ed-1-Redacted_18May2022.pdf&versionIdentifier=
- See also: D6070C00004 CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6070C00004&attachmentIdentifier=ffb0494a-509e-4883-9486-10075daf7ef7&fileName=d6070c00004-study-synopsis-Redacted_18May2022.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results data are reported per the primary completion date. There will be no updated results for all outcome measures at the time of end of study.
Groups:
- Oleclumab Dose 1 + Osimertinib Dose 1: In Part 1 (dose-escalation), participants received intravenous oleclumab (MEDI9447) Dose 1 every 2 weeks (Q2W) and oral osimertinib Dose 1 once daily (QD).
- Oleclumab Dose 2 + Osimertinib Dose 1: In Part 1 (dose-escalation), participants received intravenous oleclumab Dose 2 Q2W and oral osimertinib Dose 1 QD. In Part 2 (dose-expansion), participants (including participants dosed at the RP2D in Part 1) received IV oleclumab Dose 2 Q2W and oral osimertinib Dose 1 QD until documentation of disease progression, intolerable toxicity, or development of other reason for treatment discontinuation, whichever occurred first.
- Oleclumab Dose 1 + AZD4635 Dose 1: In Part 1 (dose-escalation), participants received intravenous oleclumab Dose 1 Q2W and oral AZD4635 Dose 1 QD.
- Oleclumab Dose 1 + AZD4635 Dose 2: In Part 1 (dose-escalation), participants received intravenous oleclumab Dose 1 Q2W and oral AZD4635 Dose 2 QD.
- Oleclumab Dose 2 + AZD4635 Dose 2: In Part 1 (dose-escalation), participants received intravenous oleclumab Dose 2 Q2W and oral AZD4635 Dose 2 QD.
Period: Overall Study
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Started | 5 | 21 | 6 | 6 | 5
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 21 | 6 | 6 | 5
Not completed — Death | 2 | 9 | 3 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 1 | 0
Not completed — Other | 1 | 11 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2 | Total
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (2.9) | 61.4 (10.3) | 64.5 (10.3) | 65.2 (13.1) | 70.6 (8.8) | 63.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 4 | 5 | 4 | 27
  Male | 1 | 11 | 2 | 1 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 21 | 6 | 6 | 5 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 19 | 0 | 2 | 1 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 6 | 4 | 4 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) in Part 1
Description: A DLT was defined as >= Grade 3 toxicity or adverse events (AE) occurred during DLT evaluation period which included any Grade 4 immune-mediated (immune nature) AE, anemia, thrombocytopenia (present > 4 days), or neutropenia (present > 4 days); >= Grade 3 colitis or pneumonitis or interstitial lung disease (ILD); >= Grade 3 nausea, vomiting, or diarrhea (not resolved to <= Grade 2 in 3 days); Grade 2 pneumonitis or ILD (not resolved to <= Grade 1 in 3 days); Grade 3 thrombocytopenia with bleeding, any grade febrile neutropenia; convulsions, seizures, or stroke; protocol defined elevations of isolated liver transaminase, isolated total bilirubin (TBL), or Hy's Law; confirmed QT interval corrected for heart rate by Fridericia's formula prolongation (>= 501 msec) on triplicate electrocardiograms within a short period of time; or any other toxicity greater than that at baseline, was clinically significant and/or unacceptable, and was judged to be a DLT by the Dose Escalation Committee.
Time Frame: From Day 1 to Day 28 after first dose of study drug
Population: The DLT-evaluable population included all participants who enrolled in the dose-escalation phase, received all planned doses of oleclumab and at least 75% of the daily administrations of osimertinib or AZD4635 during the DLT-evaluation period and completed the safety follow-up through the DLT-evaluation period or experienced any DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 3 | 4 | 3 | 5 | 4
Participants | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) in Parts 1 and 2
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Participants
  Any TEAEs | 5 | 21 | 6 | 5 | 5
  Any TESAEs | 3 | 6 | 4 | 1 | 3

3. Primary Outcome: Number of Participants With Abnormal Laboratory Parameters Reported as TEAEs in Parts 1 and 2
Description: Participants with abnormal laboratory parameters reported as TEAEs are reported. Laboratory analysis included hematology, clinical chemistry, thyroid function tests, and urinalysis.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Participants
  Anaemia | 2 | 0 | 1 | 1 | 0
  Neutropenia | 1 | 1 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 2 | 0 | 0 | 0
  Amylase increased | 1 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 3 | 0 | 0 | 0
  Blood alkaline phosphatase increased | 0 | 2 | 0 | 0 | 0
  Blood creatinine increased | 1 | 0 | 0 | 0 | 0
  Lipase increased | 1 | 0 | 0 | 0 | 0
  Hypercholesterolaemia | 0 | 1 | 0 | 0 | 0
  Hyperglycaemia | 0 | 1 | 0 | 0 | 0
  Hyperkalaemia | 1 | 1 | 0 | 0 | 0
  Hypoalbuminaemia | 1 | 0 | 1 | 0 | 0
  Hypocalcaemia | 1 | 1 | 0 | 1 | 1
  Hypokalaemia | 1 | 1 | 0 | 0 | 0
  Hypomagnesaemia | 0 | 1 | 0 | 0 | 0
  Hyponatraemia | 1 | 1 | 1 | 0 | 0
  Hypophosphataemia | 1 | 0 | 0 | 0 | 0
  Leukopenia | 0 | 0 | 0 | 1 | 0
  Blood albumin decreased | 0 | 0 | 0 | 0 | 1
  Haemoglobin decreased | 0 | 0 | 1 | 0 | 0
  Neutrophil count decreased | 0 | 2 | 0 | 1 | 0
  White blood cell count decreased | 0 | 0 | 0 | 1 | 0
  Hypercalcaemia | 0 | 0 | 1 | 0 | 0
  Thrombocytopenia | 0 | 1 | 0 | 0 | 0
  Hypothyroidism | 0 | 1 | 0 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 1 | 0 | 0 | 0
  Platelet count decreased | 0 | 2 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Vital Signs and Physical Examination Reported as TEAEs in Parts 1 and 2
Description: Participants with abnormal vital signs (heart rate, blood pressure, temperature, and respiratory rate) and physical examination reported as TEAEs are reported.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Participants
  Hypertension | 1 | 0 | 0 | 0 | 0
  Hypotension | 1 | 0 | 0 | 0 | 0
  Pyrexia | 0 | 1 | 0 | 0 | 0
  Hypoxia | 0 | 0 | 1 | 0 | 1

5. Primary Outcome: Number of Participants With Notable QTc Interval in Parts 1 and 2
Description: Notable QTc intervals included single beat changes from baseline (Day 1) values (> 30, > 60, and > 90 milliseconds). Participants who had notable QTc interval are reported.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Participants
  Single Beat change from baseline, Change > 30 milliseconds | 2 | 6 | 2 | 2 | 1
  Single Beat change from baseline, Change > 60 milliseconds | 0 | 2 | 0 | 0 | 0
  Single Beat change from baseline, Change > 90 milliseconds | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants With Objective Response (OR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in Part 2
Description: The OR is defined as confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline, and non-progressive disease and not evaluable or no non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oleclumab Dose 2 + Osimertinib Dose 1
Number analyzed (Participants) | 21
Percentage of participants | 19 [5.4 to 41.9]

7. Secondary Outcome: Duration of Response (DoR) Per RECIST v 1.1 for Parts 1 and 2
Description: The DoR is defined as duration from the first documentation of OR (confirmed CR or PR) to the first documented disease progression based on RECIST v1.1 guidelines or death due to any cause, whichever occurs first. A CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. A PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline, and non-progressive disease and not evaluable or no non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between. The progressive disease is defined at least a 20% increase in sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The DoR was analyzed using Kaplan-Meier method.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received. The DoR was analyzed for participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 2 | 4 | 0 | 0 | 0
Months | 11.4 [4.8 to 18.1] | NA [9.2 to NA] — Median and upper limit of 95% confidence interval (CI) were not derived due to insufficient events being observed at the time of the analysis. |  |  |

8. Secondary Outcome: Percentage of Participants With Disease Control (DC) in Parts 1 and 2
Description: The DC is defined as percentage of participants with CR, PR, or stable disease (SD, which was maintained by >= 8 week) based on RECIST v1.1 guidelines. A CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. A PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline, and non-progressive disease and not evaluable or no non-target lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum longest diameter since the study treatment started, and non-progressive disease and not evaluable or no non-target lesion.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Percentage of participants | 80.0 [28.4 to 99.5] | 81.0 [58.1 to 94.6] | 0 [NA to NA] — 95% CI was not derived due to insufficient events being observed at the time of the analysis. | 16.7 [0.4 to 64.1] | 0 [NA to NA] — 95% CI was not derived due to insufficient events being observed at the time of the analysis.

9. Secondary Outcome: Progression Free Survival (PFS) for Parts 1 and 2
Description: The PFS is defined as the time from the start of study treatment until the documentation of disease progression based on RECIST version 1.1 or death due to any cause, whichever occurs first, regardless of whether the participant received subsequent anticancer treatment prior to progression. The progressive disease is defined at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. Participants who were alive and progression-free at the time of data cut-off for analysis had PFS censored at the last tumor assessment date. The PFS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Months | 6.5 [1.4 to 19.8] | 11.0 [3.7 to NA] — Upper limit of 95% CI was not derived due to insufficient events being observed at the time of the analysis. | 1.4 [0.5 to 1.8] | 1.8 [0.8 to 5.5] | 1.9 [1.4 to 2.3]

10. Secondary Outcome: Overall Survival (OS) for Parts 1 and 2
Description: The OS is defined as the time from the start of study treatment until death due to any cause. Participants who are alive at the time of data cut-off had OS censored at the last known to be alive date. The OS was estimated using Kaplan-Meier method.
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Months | 21.9 [1.4 to NA] — Upper limit of 95% CI was not derived due to insufficient events being observed at the time of the analysis. | 24.8 [12.3 to NA] — Upper limit of 95% CI was not derived due to insufficient events being observed at the time of the analysis. | 16.4 [1.0 to 16.4] | 27.4 [1.5 to NA] — Upper limit of 95% CI was not derived due to insufficient events being observed at the time of the analysis. | 7.1 [1.9 to NA] — Upper limit of 95% CI was not derived due to insufficient events being observed at the time of the analysis.

11. Secondary Outcome: Percentage of Participants With OR by T790M Status at Baseline (Determined by a Central Laboratory) for Parts 1 and 2
Description: The T790M status was determined by plasma testing in a central laboratory at Baseline (Days -28 to -1). The OR is defined as confirmed CR or confirmed PR based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline, and non-progressive disease and not evaluable or no non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between. Cell-free circulating tumor deoxyribonucleic acid (ctDNA) from liquid biopsy was used as a surrogate marker for T790M status in tumor tissue.
Time Frame: From Baseline (Days -28 to -1) through 90 days of the last dose of study drug (approximately 37 months)
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received. 'Number of participants analyzed' denotes participants who had T790M status positive or negative at baseline (Days -28 to -1). The T790M status results was assessed only for participants in 'Oleclumab + Osimertinib' arms.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1
Number analyzed (Participants) | 5 | 20
Percentage of participants
  OR by T790M status positive: number analyzed (Participants) | 1 | 3
  OR by T790M status positive | 100 [2.5 to 100] | 66.7 [9.4 to 99.2]
  OR by T790M status negative: number analyzed (Participants) | 4 | 17
  OR by T790M status negative | 25.0 [0.6 to 80.6] | 11.8 [1.5 to 36.4]

12. Secondary Outcome: Percentage of Participants With DC by T790M Status at Baseline (Determined by a Central Laboratory) for Parts 1 and 2
Description: The T790M status was determined by plasma testing in a central laboratory at Baseline (Days -28 to -1). The DC is defined as percentage of participants with CR, PR, or SD (maintained by >= 8 week) based on RECIST v1.1 guidelines. A CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. A PR is defined as >= 30% decrease in the sum of longest diameters of target lesions compared to baseline, and non-progressive disease and not evaluable or no non-target lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum longest diameter since the study treatment started, and persistence of one or more non-target lesion(s). Cell-free circulating tumor deoxyribonucleic acid (ctDNA) from liquid biopsy was used as a surrogate marker for T790M status in tumor tissue.
Time Frame: From Baseline (Days -28 to -1) through 90 days of the last dose of study drug (approximately 37 months)
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received. 'Number of participants analyzed' denotes participants who had T790M status positive or negative at baseline (Days -28 to -1).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1
Number analyzed (Participants) | 5 | 20
Percentage of participants
  DC by T790M status positive: number analyzed (Participants) | 1 | 3
  DC by T790M status positive | 100 [2.5 to 100] | 100 [29.2 to 100]
  DC by T790M status negative: number analyzed (Participants) | 4 | 17
  DC by T790M status negative | 75.0 [19.4 to 99.4] | 82.4 [56.6 to 96.2]

13. Secondary Outcome: Observed Serum Concentration at the Time of End of Infusion (CEOI) of Oleclumab (MEDI9447) Over Time
Description: The CEOI of oleclumab is reported.
Time Frame: Predose (within 90 minutes prior to start of infusion) and postdose (10 minutes after the end of infusion) on Days 1 and 57
Population: Pharmacokinetic (PK) population included all participants who received any study drug, analyzed according to the treatment they actually received, and had at least one quantifiable post-dose concentration with no important protocol deviations or AEs considered to impact the PK data. 'Number of participants analyzed' denotes the number of participants evaluated for this outcome measure. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 5 | 6 | 3
µg/mL
  Day 1 | 545.7 (22.29) | 787.6 (31.27) | 494.6 (23.69) | 385.4 (23.51) | 633.3 (33.45)
  Day 57: number analyzed (Participants) | 3 | 16 | 0 | 1 | 2
  Day 57 | 926.4 (15.55) | 1183 (24.76) |  | NA (NA) — Geometric mean and geometric coefficient of variation (CV) were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point.

14. Secondary Outcome: Observed Lowest Serum Concentration (Ctrough) of MEDI9447 Over Time
Description: The Ctrough of oleclumab is reported.
Time Frame: Predose (within 90 minutes prior to start of infusion) on Day 57
Population: The PK population included all participants who received any study drug, analyzed according to the treatment they actually received, and had at least one quantifiable post-dose concentration with no important protocol deviations or AEs considered to impact the PK data. ''Number of participants analyzed' denotes the number of participants who had adequate PK sample and were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 3 | 18 | 0 | 2 | 2
µg/mL | 271.5 (38.03) | 315.5 (35.42) |  | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point.

15. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Osimertinib and Its Metabolite (AZ5104)
Description: The Cmax of osimertinib and AZ5104 are reported.
Time Frame: Predose (within 90 minutes prior to start of infusion) and postdose (1, 2, and 4 hours) on Days 1 and 29
Population: The PK population included all participants who received any study drug, analyzed according to the treatment they actually received, and had at least one quantifiable post-dose concentration with no important protocol deviations or AEs considered to impact the PK data. 'Number of participants analyzed' denotes the number of participants evaluated for this outcome measure. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1
Number analyzed (Participants) | 5 | 21
nM
  Osimertinib, Day 1: number analyzed (Participants) | 4 | 20
  Osimertinib, Day 1 | 151.9 (18.73) | 130.5 (92.63)
  Osimertinib, Day 29: number analyzed (Participants) | 3 | 20
  Osimertinib, Day 29 | 529.9 (28.46) | 484.9 (48.69)
  AZ5104, Day 1: number analyzed (Participants) | 4 | 19
  AZ5104, Day 1 | 3.271 (60.73) | 3.954 (72.97)
  AZ5104, Day 29: number analyzed (Participants) | 3 | 20
  AZ5104, Day 29 | 52.06 (43.62) | 45.30 (53.84)

16. Secondary Outcome: Cmax of AZD4635 and Its Metabolites (SSP-005173X and SSP-005174X)
Description: The Cmax of AZD4635, SSP-005173X, and SSP-005174X are reported.
Time Frame: Predose (within 90 minutes prior to start of infusion) and postdose (1, 2, 4, 6, and 24 hours) on Days 1 and 57
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 6 | 6 | 3
ng/mL
  AZD4635, Day 1 | 548.2 (19.57) | 330.6 (34.02) | 319.5 (17.93)
  AZD4635, Day 57: number analyzed (Participants) | 0 | 1 | 2
  AZD4635, Day 57 |  | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were no derived due to insufficient observations (n<3) at the specified time point.
  SSP-005173X, Day 1 | 9.238 (62.78) | 12.54 (52.36) | 6.747 (66.91)
  SSP-005173X, Day 57: number analyzed (Participants) | 0 | 1 | 2
  SSP-005173X, Day 57 |  | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point.
  SSP-005174X, Day 1 | 67.78 (30.28) | 58.18 (54.66) | 40.60 (32.19)
  SSP-005174X, Day 57: number analyzed (Participants) | 0 | 1 | 2
  SSP-005174X, Day 57 |  | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point.

17. Secondary Outcome: Tmax of AZD4635 and Its Metabolites (SSP-005173X and SSP-005174X)
Description: The Tmax of AZD4635, SSP-005173X, and SSP-005174X are reported.
Time Frame: Predose (within 90 minutes prior to start of infusion) and postdose (1, 2, 4, 6, and 24 hours) on Days 1 and 57
Population: as for outcome 15
Measure: Median (Full Range); unit: Hour
Arm/Group | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 6 | 6 | 3
Hour
  AZD4635, Day 1 | 1.03 [1.00 to 2.13] | 1.07 [1.00 to 1.08] | 1.05 [1.02 to 1.22]
  AZD4635, Day 57: number analyzed (Participants) | 0 | 1 | 2
  AZD4635, Day 57 |  | NA [NA to 2.13] — Median and upper limit of range were not derived due to insufficient observations (n<3) at the specified time point. | NA [0.917 to 1.00] — Median was not derived due to insufficient observations (n<3) at the specified time point.
  SSP-005173X, Day 1 | 1.54 [1.00 to 2.13] | 1.93 [1.02 to 2.03] | 1.22 [1.02 to 2.07]
  SSP-005173X, Day 57: number analyzed (Participants) | 0 | 1 | 2
  SSP-005173X, Day 57 |  | NA [NA to 2.13] — Median and lower limit of range were not derived due to insufficient observations (n<3) at the specified time point. | NA [0.917 to 1.00] — Median was not derived due to insufficient observations (n<3) at the specified time point.
  SSP-005174X, Day 1 | 1.03 [1.00 to 2.13] | 1.07 [1.00 to 1.87] | 1.05 [1.02 to 1.22]
  SSP-005174X, Day 57: number analyzed (Participants) | 0 | 1 | 2
  SSP-005174X, Day 57 |  | NA [NA to 2.13] — Median and lower limit of range were not derived due to insufficient observations (n<3) at the specified time point. | NA [NA to 1.00] — Median and lower limit of range were not derived due to insufficient observations (n<3) at the specified time point.

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) of AZD4635 and Its Metabolites (SSP-005173X and SSP-005174X)
Description: The AUC0-24 of AZD4635, SSP-005173X, and SSP-005174X are reported.
Time Frame: Predose (within 90 minutes prior to start of infusion) and postdose (1, 2, 4, 6, and 24 hours) on Days 1 and 57
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 6 | 6 | 3
h*ng/mL
  AZD4635, Day 1: number analyzed (Participants) | 5 | 4 | 3
  AZD4635, Day 1 | 2546 (27.24) | 1324 (28.02) | 1624 (20.32)
  AZD4635, Day 57: number analyzed (Participants) | 0 | 1 | 2
  AZD4635, Day 57 |  | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point.
  SSP-005173X, Day 1: number analyzed (Participants) | 4 | 5 | 3
  SSP-005173X, Day 1 | 84.08 (94.72) | 76.57 (68.17) | 59.88 (61.87)
  SSP-005173X, Day 57: number analyzed (Participants) | 0 | 1 | 2
  SSP-005173X, Day 57 |  | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point.
  SSP-005174X, Day 1: number analyzed (Participants) | 5 | 5 | 3
  SSP-005174X, Day 1 | 304.4 (54.74) | 231.9 (65.94) | 192.4 (24.54)
  SSP-005174X, Day 57: number analyzed (Participants) | 0 | 1 | 2
  SSP-005174X, Day 57 |  | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point. | NA (NA) — Geometric mean and geometric CV were not derived due to insufficient observations (n<3) at the specified time point.

19. Secondary Outcome: Number of Participants With Positive Post-baseline for Anti-oleclumab Antibodies
Description: Number of participants with positive post-baseline for anti-oleclumab antibodies are reported.
Time Frame: Predose on Days 1 (Baseline), 29, and 57, and later every 12 weeks through the 12 months and 90 days after the last dose of study drug (approximately 37 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
Number analyzed (Participants) | 5 | 21 | 6 | 6 | 5
Participants | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 through 90 days of the last dose of study drug (approximately 37 months)
Arm/Group | Oleclumab Dose 1 + Osimertinib Dose 1 | Oleclumab Dose 2 + Osimertinib Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 1 | Oleclumab Dose 1 + AZD4635 Dose 2 | Oleclumab Dose 2 + AZD4635 Dose 2
All-Cause Mortality (participants affected / at risk) | 2/5 | 9/21 | 3/6 | 2/6 | 3/5
Serious Adverse Events (participants affected / at risk) | 3/5 | 6/21 | 4/6 | 1/6 | 3/5
Other Adverse Events (participants affected / at risk) | 5/5 | 21/21 | 6/6 | 5/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oleclumab Dose 1 + Osimertinib Dose 1 (N=5) | Oleclumab Dose 2 + Osimertinib Dose 1 (N=21) | Oleclumab Dose 1 + AZD4635 Dose 1 (N=6) | Oleclumab Dose 1 + AZD4635 Dose 2 (N=6) | Oleclumab Dose 2 + AZD4635 Dose 2 (N=5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oleclumab Dose 1 + Osimertinib Dose 1 (N=5) | Oleclumab Dose 2 + Osimertinib Dose 1 (N=21) | Oleclumab Dose 1 + AZD4635 Dose 1 (N=6) | Oleclumab Dose 1 + AZD4635 Dose 2 (N=6) | Oleclumab Dose 2 + AZD4635 Dose 2 (N=5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (11) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (7) | 4 (6) | 3 (3) | 2 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (4) | 5 (6) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 3 (3) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (5) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual brightness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Arm B (Oleclumab + AZD4635 groups) did not proceed to the dose expansion phase due to lack of response to treatment and a change in the formulation of AZD4635. The OR and DC by T790M status for 'Oleclumab + AZD4635' groups were not conducted due to the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03381274/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03381274/SAP_001.pdf